CLINICAL TRIAL: NCT01208376
Title: Prevalence of Liver Fibrosis and Progression of Liver Fibrosis in HIV-infected, Hepatitis C (HCV) and Hepatitis B (HBV) Seronegative Patients With Chronic Alanine Aminotransferase (ALT) Elevation
Brief Title: Prevalence of Liver Fibrosis and Progression of Liver Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Helen Kovari-Kramer (Other)
Collaborators: Swiss HIV Cohort Study (Network)
Responsible Party: Sponsor-Investigator, Helen Kovari-Kramer, MD, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: SHCS 625
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-05

CONDITIONS: HIV Infection and Chronic Alanine Aminotransferase Elevation
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- unexplained chronic ALT elevation: Case patients: HIV-infected, unexplained chronic alanine aminotransferase (ALT) elevation
  Interventions: Other: Fibroscan
- always normal ALT: Control patients: HIV-infected, always normal ALT values
  Interventions: Other: Fibroscan

INTERVENTIONS:
Other: Fibroscan — Fibroscan and Serum Fibrose-marker
  Other Names: Fibroscan and Serum Fibrose-marker

SUMMARY:
Little is known about the clinical significance of chronic alanine aminotransferase (ALT) elevation in HIV-infected patients without hepatitis B and C coinfection. Study aim is first to evaluate the prevalence of liver fibrosis and cirrhosis in HIV-infected patients with chronic ALT elevation and no chronic viral hepatitis using non-invasive diagnostic tests and second to find associated factors with significant fibrosis and cirrhosis. In a second longitudinal part we intend to assess fibrosis progression within 1 and 3 years.

ELIGIBILITY:
Inclusion criteria: Case patients:

* HIV-1 infection
* no hepatitis B and C coinfection
* chronic alanine aminotransferase (ALT) elevation after 1.1.2007
* signed informed consent
* no other common cause of liver disease

Control patients:

* HIV-infection
* no hepatitis B and C coinfection
* no ALT elevation after 1.1.2002, the date when ALT values were regularly collected in the Swiss HIV Cohort Study (SHCS)
* no known chronic liver disease

Exclusion criteria: please see inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected, hepatitis B and C seronegative Patients With Chronic alanine aminotransferase (ALT) Elevation
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2010-10; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Liverfibrosis | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland